CLINICAL TRIAL: NCT04553146
Title: Immediate Implant Placement in the Posterior Region Combining Socket Seal Abutment and Alveolar Ridge Preservation: Implant, Hard and Soft Tissue Outcomes After 1 Year, 3 Years and 5 Years
Brief Title: Clinical and Dimensional Outcomes of Sealing Socket Abutment Combined to Alveolar Ridge Preservation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Liege (Other)
Collaborators: Institut Straumann AG (Industry)
Responsible Party: Principal Investigator, Dr. France LAMBERT, Head and Chair of Department, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2017-BLX
Record Dates: First submitted 2020-09-04; First posted 2020-09-17 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Non-maintainable Posterior Tooth (Molars and Premolars)
MeSH Terms: conditions — Bicuspid Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): immediate implant placement in posterior sites using a custom-made sealing socket abutment combined to alveolar ridge preservation
  Interventions: Procedure: Immediate implantation in posterior region with alveolar ridge preservation combined with sealing socket abutment

INTERVENTIONS:
Procedure: Immediate implantation in posterior region with alveolar ridge preservation combined with sealing socket abutment — Twenty BLXⓇ Straumann immediate implants were placed flapless. The gap around the implant was filled with xenogeneic biomaterial. An intra-oral scanner was performed and sent to the dental laboratory to digitally design a customized healing abutment. The abutment was then milled from a block of PEEK and placed a couple of hours later in the clinic. Three months after implantation, the abutment was removed and the final monolithic crown based on the initial IOS was placed. The transmucosal design from the SSA was replicated on the final crown.

SUMMARY:
objectives

The aim of this study was to assess the implant outcomes as well as hard and soft tissue dimensional changes of immediate implant placement in posterior sites using a custom-made sealing socket abutment (SSA) combined to alveolar ridge preservation (ARP).

Material and methods

Twenty posterior teeth were immediately replaced with implants in 20 patients. The remaining sockets were filled with Deproteinized Bovine Bone Mineral. Based on intra-oral scanners (IOS), custom-made SSAs were placed the same day. CBCT and IOS were performed to monitor hard and soft tissue dimensional changes. Moreover, implant survival rate, peri-implant bone changes, peri-implant health and pink esthetic score were recorded at 1 year, 3years and 5 years.

DETAILED DESCRIPTION:
Study population

Hopeless maxillary or mandibular molars with tooth anatomy and bone anchorage allowing an immediate implant procedure: apical bone height of at least 5 mm or presence of interradicular septum, socket with intact bone walls, absence a large apical periodontitis, Patients needing tooth replacement in the posterior region (molars) will be recruited from the Department of Periodontology and Oral and Implant Surgery of the University of Liège, Belgium.

Procedures

After a local anesthesia, one of the two experienced surgeons (LF or LG) proceeded to the least traumatic extraction of the concerned tooth. The consecutive drills for implant placement were carried out while considering the future position of the crown for a screw- retained restoration. Twenty BLX implants (Roxolid®, SLAactive®, Institut Straumann AG) were placed flapless with a sufficient apical or septum anchorage and the insertion torque was recorded. The gap around the implant was filled with deproteinized bovine bone mineral (DBBM) (cerabone®, botiss biomaterials GmbH).

Just after the implant placement, an intra-oral scan (IOS) (Trios 3®, 3-Shape) with a scanbody connected onto the implant platform was performed and sent to the dental laboratory to digitally design (Dental Wings®) a customized healing abutment. The SSA was then milled (CARES®, Institut Straumann AG) from a block of PEEK (JUVORATMPEEK, JUVORATM Ltd. National Distributor: Institut Straumann AG), cemented to a titanium abutment (Variobase®, Institut Straumann AG) and provided to the patient on the same day. During manufacturing of the SSA, a conventional healing abutment was screwed on the implant and a collagen sponge (Collaplug®) was provisionally placed buccally to protect the exposed biomaterial until the placement of the SSA. A standardized parallel peri-apical radiograph using a custom-made film holder was taken in order to record the baseline bone level. Each patient was instructed to rinse twice daily with an aqueous solution of 0.2% chlorhexidine (Corsodyl®, GSK) and to avoid brushing of the area until the first recall 10-12 days later. Anti-inflammatories (Ibuprofen® 600 mg) and additional analgesics (Paracetamol® 500 mg) were prescribed and taken according to the patient's needs. If the surgeon deemed it necessary, an anti- biotic was prescribed (Amoxicillin® 500mg 3x/day during 5 days). Three months after implantation, the abutment was removed, the osseointegration of the implant was checked and the final lithium aluminosilicate ceramic reinforced with lithium disilicate monolithic crown (n!ce® glass-ceramic block, Institut Straumann AG) based on the initial IOS was cemented to a titanium abutment (Variobase®, Institut Straumann AG) and placed. The transmucosal design from the SSA was replicated on the final crown. Follow-up evaluations and data recording will be performed 7-10 days, 3 months, 6 months, 12 months, 3years and 5years after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* good general health (ASA I/II),
* more than 18 years old,
* non smoker,
* one hopeless tooth,
* healthy periodontal condition,
* the presence of at least 2 mm of keratinized gingiva,
* adequate plaque control (FMPS ≤ 25%), adequate bone quantity in the septum if present and at least 5 mm of bone in the apical region

Exclusion Criteria:

* auto-immune disease or immunocompromised patients,
* uncontrolled diabetes,
* use of steroids or biphosphonates,
* local or systemic infection (medical treatment needed prior to entrance to the study), pregnancy or breastfeeding, alcoholism or chronically drug abuse.

Local exclusion criteria:

* bone availability requiring an angulated abutment,
* untreated local inflammation,
* cyst,
* mucosal disease or oral lesions,
* local irradiation therapy,
* oral communication with sinus after the extraction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline to 1 year of the bone remodeling : horizontal measurements (based on CBCT, in mm) | Baseline to 1, 3 and 5 years
  The measurements were done by matching and superimposing CBCT using a three dimensional reconstruction software. The measures were performed from implant platform to 7 mm below this reference line. Bucco-palatal remodeling, buccal remodeling and palatal/lingual remodeling were measured
Changes from Baseline to 1 year of the bone remodeling : vertical measurements (based on CBCT, in mm) | Baseline to 1, 3 and 5 years
  The measurements were done by matching and superimposing CBCT using a three dimensional reconstruction software. Four vertical measurements were taken : on the buccal side, on the lingual side, and in mesial and distal of the implant, under the contact points.
Changes from baseline to 6 months and to 1 year of the soft tissue profiles (based on intra-oral scanners, in mm) | Baseline to 1, 3 and 5 years
  Intra-oral scanners were performed at baseline, 6 months and 1 year and were superimposed using a specific software. The buccal and lingual/palatal measurements were done perpendicular to the soft tissue profile at gingival margin and every mm below until 4 mm. The recession was measure as the vertical distance between the gingival margin at the different time points.

SECONDARY OUTCOMES:
implant survival rate (based on criteria of Buser et al., 1990) | Baseline to 1, 3 and 5 years
  Success was defined according to the criteria of Buser et al., 1990 which are 1. absence of suppuration (recurring peri implant infection) 2. absence of persistent complaints like pain, foreign body sensation and/or dysesthesia 3. absence of continuous radioluncency area around the implant 4. absence of implant mobility.
Pocket depth around the implant (based on probing, in mm) | Baseline to 1, 3 and 5 years
  PD was measured by means of a periodontal probe (CP 15 UNC, Hu-Friedy, Chicago, IL, USA) at 6 sites per implant and rounded off to the nearest millimeter.
Peri-implant bone level changes (based on periapical radiography, in mm) | Baseline to 1, 3 and 5 years
  The peri-implant bone levels were assessed on periapical radiography using the parallel technique: the linear distance between the implant shoulder of the bone level implants and the first bone to implant contact (DIB, mm) was measured at the mesial and distal aspects using the specific software Image J64 (National Institutes of Health, Bethesda, MD, USA). Final DIB values were recorded as the average of the obtained mesial and distal values.
Pink esthetic score (based on PES questionnaire of Furhauser et al, 2005) | Baseline to 1, 3 and 5 years
  The PES compares the peri-implant soft tissue conditions to the respective features present at the contralateral natural tooth site. A score of 0, 1 or 2 was assigned to each parameter (mesial and distal papilla, soft tissue contour, soft tissue level, alveolar process, soft tissue coloring and texture), the highest possible score being 14, as described by Fürhauser et al (Fürhauser et al., 2005).
Plaque index around the implant (based on classification of Mombelli et al, 1987) | Baseline to 1, 3 and 5 years
  The plaque index was scored according to Mombelli 1987 (0 = no detection of plaque; 1 = plaque only recognized by running a probe across the smooth marginal surface of the implant, 2 = plaque can be seen by the naked eye, 3 = abundance of soft matter)
Bleeding on Probing around the implant (based on classification of Mombelli et al, 1987) | Baseline to 1, 3 and 5 years
  The bleeding on probing was scored according to Mombelli 1987 (0 = no bleeding when a periodontal probe is passed along the gingival margin adjacent to the implant; 1 = isolated bleeding spots visible, 2 = Blood forms a confluent red line on margin, 3 = heavy or profuse bleeding)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU University of Liège, Liège, Belgium